CLINICAL TRIAL: NCT04666857
Title: Family Centred Early Intervention to Improve Motor Development of Infants With Severe Congenital Heart Disease
Brief Title: Family Centred Early Intervention of Infants With Congenital Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EMI
Record Dates: First submitted 2020-11-23; First posted 2020-12-14 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Congenital Heart Disease in Children
Keywords: congenital heart diseases; open heart surgery; motor development; early intervention; family centred; physiotherapy
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Intervention Model Description: prospective monocentric single-blinded, two-arm feasibility randomised controlled interventional pilot trial
Who Masked: Outcomes Assessor
Masking Description: Assessors will be blinded to the allocation of participants
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard care (No Intervention): Control subject will receive standard care of treatment
- intervention group (Experimental): intervention group will receive early intervention
  Interventions: Other: early motor intervention

INTERVENTIONS:
Other: early motor intervention — infants with CHD after open heart surgery will receive early intervention
  Arms: intervention group

SUMMARY:
In this study the investigators aim to test the feasibility for therapists and acceptability to parents of an early motor intervention for infants with congenital heart disease (CHD) after open heart surgery. This intervention will be compared to the standard care of treatment that is recommended for infants with congenital heart disease at the University Children Hospital Zurich.

DETAILED DESCRIPTION:
In this feasibility pilot randomised study children will be randomly assigned to a control and an intervention group. Children of the control group will receive standard of care for infants with severe CHD: cardiac surveillance, counselling and screening at the University Children's Hospital Zurich and standardised developmental checkups by their paediatrician. Physiotherapy is normally not comprised in standard of care, but some infants may receive physiotherapy, if they present with obvious signs of motor developmental delay, detected by the paediatrician later on in their life. Once enrolled in this study, an infant of the control group will not receive early motor intervention as an infant enrolled in the intervention group.

Infants randomly assigned to the intervention group will receive early motor intervention, which will be based on the results of our qualitative study. It will comprise supporting parents by a paediatric physiotherapist. Parents will be guided on how to best stimulate their infant's development during daily activities. Parents will be actively involved in the intervention with the aim to challenge their infant at the limit of its postural capacity and thus help the infant to optimize its motor repertoire. The intervention will start after baseline with infants aged 3-6 months and end after three months with infants aged 6-9 months.

The intervention will start at home, then alternating at the Children's Hospital and at home. Telephone or video counselling will be provided to support parents if needed. The order may change according to the needs of the family when necessary and adjusted to best fit the daily routine the family.

ELIGIBILITY:
Inclusion Criteria:

* Infants born with severe cyanotic and acyanotic congenital heart disease (e.g. tetralogy of Fallot, pulmonary atresia, transposition of the great arteries, atrial/ventricular septal defects, double outlet right ventricle, ...) who undergo open-heart surgery once before the first 3-6 months of their life
* Parents able to comprehend the patient information linguistically and cognitively
* Informed consent of parents as documented by signature

Exclusion Criteria:

* Infants with hypoplastic left heart syndrome as they need to undergo several open-heart surgeries within the first period of their life.
* Infants with trisomy 21 and other syndromes like 22q11 microdeletion syndrome, CHARGE syndrome that are often associated with CHD. These infants often show additional cognitive impairments that might confound the effect of our intervention.

Ages: 2 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2021-05-31 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
Dropout rate | "3 up to 6 months of age" (baseline) and at "12 months of age"
  The primary outcome will test the procedure for its acceptability, estimation the likely rates of recruitment and retention of subjects and the calculation of appropriate sample size. Further objectives are the usefulness of the outcome assessment measures.

OTHER OUTCOMES:
Hammersmith Infant Neurological Examination | "3 up to 6 months of age" (baseline) and at "12 months of age"
  The Hammersmith Infant Neurological Examination assesses different aspects of neurological function.
  the higher the scores the better, the range depends on the child's abilities metric: ordinal
General Movements | "3 up to 6 months of age" (baseline)
  The General Movement assessment is a video-based, non-invasive way to identify neurological deviations that may lead to neurodevelopmental disorders later in life.
  The more variables the motor output of infants, the better infants' neuromotor development will be.
  metric: categorial
Infant Motor Profile | "3 up to 6 months of age" (baseline), "6 up to 9 months of age" (end of intervention), at "12 months of age"
  The Infant Motor Profile is a standardised and qualitative method to assess motor behaviour in infants, a 15 minutes, video-based assessment tool, consists of 5 domains: motor variation, adaptability, symmetry, fluency and performance.
  The higher the score, the better - the range depends on the child's abilities and is age dependent metric: ordinal
Alberta Infant Motor Scale Change in being assessed at different time points at baseline, at the end of the intervention after three months and at follow up | "3 up to 6 months of age" (baseline), "6 up to 9 months of age" (end of intervention) and at "12 months of age"
  The Alberta Infant Motor Scale is an observational measure of infants' gross motor development from birth until 18 months consisting of 58 items, measuring infants' performance; The higher the score, the better, the range depends on the child's abilities and is age dependent
  metric: ordinal
Bayley Scale for Infant and Toddlers Development | "around 12 months of age"
  Bayley Scale for Infant and Toddlers Development is an internationally used and validated battery to assesses key domains of cognition, language, socio-emotional, motor and adaptive behaviour by standardized observation and rating of the play behaviour of children the higher the scores the better, the range depends on the child's abilities and is age dependent metric: ordinal
Parental Stress Index | "3 up to 6 months of age" (baseline), "6 up to 9 months of age" (end of intervention) and at "12 months of age"
  The Parental Stress Index investigates parental stress of children with all different kind of diagnoses, consists of 5 subscales assessing areas where parental strain is high; the Parental Stress Index consists of 48 items the lower, the score the better
  metric: ordinal
Brief Symptom Inventory 18 | "3 up to 6 months of age" (baseline), "6 up to 9 months of age" (end of intervention) and at "12 months of age"
  The Brief Symptom Inventory 18 contains a three six-item scales somatization, depression, and anxiety as well as the Global Severity Index the lower, the score the better
  metric: ordinal
Parental Overprotection Measure | "3 up to 6 months of age" (baseline), "6 up to 9 months of age" (end of intervention) and at "12 months of age"
  The Parental Overprotection Measure assesses parenting behaviours that restrict a child's exposure to situations containing perceived threat or harm.
  the higher the scores the more parents protect their children metric: ordinal
Family Empowerment Scale | "3 up to 6 months of age" (baseline), "6 up to 9 months of age" (end of intervention) and at "12 months of age"
  The Family Empowerment Scale measures empowerment of families. It consists of three subscales, family, service system and community/political. We use the subscale family to gather relevant information as a result of an intervention.
  the higher the scores the more the family feels empowered metric: ordinal
Quality of life form Short Form 36 | "3 up to 6 months of age" (baseline), "6 up to 9 months of age" (end of intervention) and at "12 months of age"
  The Quality of life form Short Form 36 is a widely used questionnaire assessing self-reported health related quality of life the lower the score the better
  metric: ordinal
Pediatric Quality of Life Inventory | "3 up to 6 months of age" (baseline), "6 up to 9 months of age" (end of intervention) and at "12 months of age"
  The Pediatric Quality of Life Inventory measures quality of life of infants aged 1- 24 months.
  the higher the scores the more the quality of life is affected. metric: ordinal

CONTACTS AND LOCATIONS:
Overall Officials: Bea Latal, Dr. med., Study Director — University Children's Hospital, Zurich
Locations (1):
- University Children's Hospital, Zurich, Switzerland